CLINICAL TRIAL: NCT01131962
Title: Control of Acute Variceal Bleeding Using the Multi-shooter Band Ligator Compared to Injection Sclerotherapy.
Brief Title: Comparing Two Methods to Stop Vomiting of Blood Using the Endoscope
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Yasser Hamza, Professor of Surgery, University of Alexandria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: egsbl1
Record Dates: First submitted 2010-05-26; First posted 2010-05-27 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Hematemesis; Portal Hypertension
Keywords: esophageal varices; hematemesis; endoscopy
MeSH Terms: conditions — Hematemesis; Hypertension, Portal; Esophageal and Gastric Varices

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- band ligation group (Active Comparator): this group will have immediate control of the hematemesis by endoscopic band ligation.
  Interventions: Procedure: Endoscopic control of hematemesis
- sclerotherapy group (Active Comparator): This group will have immediate control of hematemesis by endoscopic sclerotherapy
  Interventions: Procedure: Endoscopic control of hematemesis

INTERVENTIONS:
Procedure: Endoscopic control of hematemesis — Endoscopy is performed to diagnose the cause of hematemesis and to control it using band ligation or sclerotherapy
  Other Names: Six shooter band ligator; Ehanolamine oleate sclerosant material

SUMMARY:
Band ligation and injection sclerotherapy are two modalities of treatment that are applied using the endoscope. The purpose of this study is to determine which of two methods is better for controlling bleeding from the upper gut.

DETAILED DESCRIPTION:
The use of band ligation for endoscopy during the attack of hematemesis is a novel practice as opposed to injection sclerotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Active hematemesis
* esophageal varices

Exclusion Criteria:

* Hemodynamic unstability
* Hepatic coma or precoma
* Tense ascitis
* Coagulopathies
* concomitant gastric varices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-05; Primary Completion 2011-09 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
control of hematemesis | 72 hours
  Success for either techniques to be able to stop the bleeding promptly and maintain that for 72 hours

SECONDARY OUTCOMES:
occurence of complications from the intervention | 30 days
  the study subjects are reveiwed in 30 days to detect any complications secondary to the endoscopic intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Hamza, A Prof, Principal Investigator — University of Alexandria
Locations (1):
- Hematemesis unit, Alexandria Main University Hospital, Azarita, Alexandria, Egypt